CLINICAL TRIAL: NCT03539458
Title: Feasibility Study of the Tendyne Mitral Valve System for Use in Subjects With Mitral Annular Calcification
Brief Title: Feasibility Study of the Tendyne Mitral Valve System in Mitral Annular Calcification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0005-P
Record Dates: First submitted 2018-04-12; First posted 2018-05-29 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency; Mitral Annular Calcification; Mitral Annulus Calcification; Cardiovascular Diseases; Valve Heart Disease; Heart Valve Diseases; Heart Valve Calcification; Mitral Valve Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Cardiovascular Diseases; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Device Arm (Experimental): All subjects will undergo procedure with the Tendyne Mitral Valve System.
  Interventions: Device: Tendyne Mitral Valve System

INTERVENTIONS:
Device: Tendyne Mitral Valve System — Mitral valve replacement

SUMMARY:
This study is a prospective, single-arm, multi-center feasibility clinical study of the Tendyne Mitral Valve System for the treatment of eligible subjects with symptomatic, severe mitral regurgitation and severe mitral annular calcification (MAC). Subjects satisfying the study inclusion/exclusion criteria will undergo a procedure to implant the Tendyne mitral valve replacement device.

ELIGIBILITY:
Inclusion criteria:

1. Heart Team determines subject is not a suitable candidate for conventional surgical treatment due to degree of MAC present and the subject will likely benefit from transcatheter valve implantation
2. Symptomatic, severe mitral regurgitation, as defined in the 2017 ACC expert Consensus Decision Pathway on the Management of MR
3. NYHA Functional Classification ≥ II (if Class IV, patient must be ambulatory)
4. Age 18 years or older at time of consent
5. Not a member of a vulnerable population per the investigator's judgment
6. The subject or the subject's legal representative has been informed of the nature of the study and agrees to its provisions, including complying with study required testing and follow-up visits, and has provided written informed consent

Exclusion criteria:

1. Presence of Left Ventricle or Left Atrium thrombus
2. Chest condition that prevents transapical access
3. Left Ventricular Ejection Fraction (LVEF) less than 25% assessed by echocardiogram
4. Left Ventricular End Diastolic Dimension (LVEDD) > 7.0 cm
5. Severe mitral stenosis not amenable to balloon valvuloplasty or transcatheter therapy
6. Prior intervention with permanently implanted mitral device (e.g. MitraClip)
7. Mitral pathoanatomy and Left Ventricular Outflow tract (LVOT) anatomy deemed not suitable for Tendyne mitral valve implantation
8. Any planned cardiac surgery or intervention that is 30 days prior and 30 days post that is not concomitant with the Tendyne procedure
9. Cardiac resynchronization therapy (CRT) device or implantable pulse generator (IPG) implanted within three months of planned implant procedure
10. Myocardial Infarction (MI) within 30 days of the planned implant procedure
11. Symptomatic, or ischemia-associated coronary artery disease (e.g., active ischemia) amenable to revascularization and thus requiring stenting or CABG
12. Cerebrovascular accident (CVA) within six months of planned implant procedure
13. Unresolved severe symptomatic carotid stenosis (> 70% by ultrasound)
14. Cardiogenic shock or hemodynamic instability requiring inotropes or mechanical support devices within 1 month prior to planned implant procedure
15. Severe tricuspid regurgitation or severe right ventricular dysfunction
16. Hypertrophic or restrictive cardiomyopathy, constrictive pericarditis or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
17. Any of the following: leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy if cannot be adequately treated
18. History of endocarditis within 6 months of planned implant procedure
19. Active systemic infection requiring antibiotic therapy
20. Known hypersensitivity or contraindication to procedural or post-procedural medications (e.g., contrast solution, anti-coagulation therapy) which cannot be adequately managed medically
21. Subject unable or unwilling to take anticoagulation with warfarin for a minimum of 6 months following Tendyne valve implantation
22. Known hypersensitivity to nickel or titanium
23. Subject is undergoing hemodialysis due to chronic renal failure ( ≥ Stage 4 CKD)
24. Subject has pulmonary arterial hypertension (fixed PAS >70mmHg)
25. FEV1 < 50% of predicted or < 1L
26. Subject refuses blood transfusions
27. Subject has COPD requiring continuous home oxygen therapy or chronic outpatient oral steroid use
28. Pregnant, lactating, or planning pregnancy within next 12 months.
29. Currently participating in an investigational drug or another device trial that has not reached its primary endpoint
30. Subjects with non-cardiac co-morbidities that are likely to result in a life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sorajja, MD, Principal Investigator — Minneapolis Heart Institute - Abbott Northwestern Hospital; Vinod Thourani, MD, Principal Investigator — Piedmont Heart Hospital
Locations (4):
- United States (4):
  - Emory University Hospital, Atlanta, Georgia
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initially designed to register up to 30 patients from 10 investigational sites in the U.S. However only 11 patients were actually registered and underwent successful implantation with Tendyne TMVI device. Of the 11 patients, 10 patients completed 30-day follow-up, while the remaining one patient died 18 days after the implant procedure
Groups:
- Device Arm: All subjects will undergo a procedure with the Tendyne Mitral Valve System: Mitral valve replacement
Period: Overall Study
Arm/Group | Device Arm
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Device Arm
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.2 (5.8)
Age, Customized [Number; unit: participants]
  18-75 years | 4
  >75 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 1
  Not Hispanic/Latino | 10
  White/Caucasian | 10
Region of Enrollment [Number; unit: participants]
  United States | 11
Predicted Surgical Mortality [Mean (Standard Deviation); unit: Probability percentage] — The Society of Thoracic Surgeons' risk model predict the risk of operative mortality & morbidity after adult cardiac surgery. Risk models were developed for nine specific endpoints, including operative mortality. Operative mortality includes both (1) all deaths occurring during the hospitalization, even if after 30 days (2) deaths occurring after discharge, but within 30 days of the procedure. Therefore, a patient's mortality risk score is defined as the patient's predicted risk of operative mortality as calculated by the specific operative mortality statistical model.
  Probability percentage | 9.03 (8.09)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (5.9)
Renal Insufficiency (GFR < 60 mL/min/1.73m^2) [Count of Participants; unit: Participants] | 5
Peripheral Artery Disease [Count of Participants; unit: Participants] | 6
History of Hypertension [Count of Participants; unit: Participants] | 10
Coronary Artery Disease [Count of Participants; unit: Participants] | 8
Prior Coronary Intervention [Count of Participants; unit: Participants] | 8
Previous Myocardial Infarction [Count of Participants; unit: Participants] | 3
Prior Valve Intervention [Count of Participants; unit: Participants] | 6
LV Measurement [Mean (Standard Deviation); unit: mL]
  Left Ventricular End Diastolic Volume (LVEDV) | 117.3 (27.1)
  Left Ventricular End Systolic Volume (LVESV) | 48.7 (18.4)
LV Measurement [Mean (Standard Deviation); unit: cm]
  Left Ventricular End Diastolic Diameter (LVEDD) | 5.2 (0.4)
  Left Ventricular End Systolic Diameter (LVESD) | 3.7 (0.6)
Kansas City Cardiovascular Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL) within a 2-week recall period. Scores are scaled 0-100, where a score of 100 represents the lowest burden of symptoms.
  units on a scale | 46.0 (20.1)
NYHA Functional Class [Number; unit: participants] — Class I: Patients with cardiac disease but without resulting limitations of physical activity. Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Class III: Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or anginal syndrome may be present even at rest & discomfort is increased with physical activity.
  participants
    NYHA Functional Class I | 0
    NYHA Functional Class II | 2
    NYHA Functional Class III | 9
    NYHA Functional Class IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Endpoint of Device Success and Freedom From Device or Procedure Related Serious Adverse Events (SAEs), as Classified by the Clinical Events Committee (CEC)
Description: Definition of Device Success:
  All of the following must be present:
  1. Absence of procedural mortality or stroke; and
  2. Proper placement and positioning of the device, and
  3. Freedom from unplanned surgical or interventional procedures related to the device or access procedure; and
  4. Continued intended safety and performance of the device, including:
  i. No evidence of structural or functional failure
  ii. No specific device-related technical failure issues or complications
  iii. Reduction of MR to either optimal or acceptable levels without significant structural valve dysfunction and with no greater than mild (1+) paravalvular MR (and without associated hemolysis).
  All device- or procedure-related adverse events will be adjudicated by an independent clinical events committee
Time Frame: 30 days post implant
Population: The number of participants analyzed includes all subjects that were registered and implanted in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Arm
Number analyzed (Participants) | 11
Participants | 7

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Device Arm
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device Arm (N=11)
Bleeding (Blood and lymphatic system disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 1
Paravalvular Leak (Blood and lymphatic system disorders) | 1
Arrhythmia or conduction disturbance (Cardiac disorders) | 1
Worsening Congestive Heart Failure (Cardiac disorders) | 1
Mesenteric Ischemia and Hemorrhagic Shock (Gastrointestinal disorders) | 1
Stroke/TIA (Nervous system disorders) | 1
Respiratory insufficiency/Failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Device Arm (N=11)
Bleeding (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Arrhythmia or Conduction Disturbance (Cardiac disorders) | 2
Heart Failure treated with IV diuretics (Cardiac disorders) | 1
Vocal Cord Dysfunction (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Dizziness (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not use study-related data without the written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT03539458/Prot_SAP_000.pdf